CLINICAL TRIAL: NCT05759611
Title: Definition of Respiratory Training Protocols in Obese Patients
Brief Title: Definition of Respiratory Training Protocols in Obese Patients (PROALRESPIOB)
Acronym: PROALRESPIOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01C024
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Obesity
Keywords: Obesity; Respiratory training; Rehabilitation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (CTRL) (Other)
  Interventions: Other: Standard integrated metabolic rehabilitation protocol + guided spontaneous breathing exercises
- Experimental group (RMT) (Experimental)
  Interventions: Other: Standard integrated metabolic rehabilitation protocol + specific respiratory muscle training program

INTERVENTIONS:
Other: Standard integrated metabolic rehabilitation protocol + guided spontaneous breathing exercises — Physical exercise protocol before and after 12 sessions of standard integrated metabolic rehabilitation protocol + guided spontaneous breathing exercises lasting about 20 minutes per session
  Arms: Control group (CTRL)
Other: Standard integrated metabolic rehabilitation protocol + specific respiratory muscle training program — Physical exercise protocol before and after 12 sessions of standard integrated metabolic rehabilitation protocol + a specific respiratory muscle training program according to the protocol recently proposed by Spengler et al. (Wuthrich et al., 2015; Schaer et al., 2018), adapted according to the baseline characteristics of the respiratory function of the subjects.
  Arms: Experimental group (RMT)

SUMMARY:
The project is aimed at investigating the effectiveness of respiratory training protocols in relieving exercise dyspnea, improving respiratory efficiency and the ability to perform physical activity, even daily, in obese patients.

Therefore, some respiratory exercises with different characteristics and mechanisms of action will be introduced into the standard program of integrated metabolic rehabilitation implemented at the Istituto Auxologico Italiano, Piancavallo, Italy (Division of Auxology and Division of Metabolic Diseases) in order to identify a suitable training protocol for this population, the development of which can be carried out over time by patients even autonomously (Sheel and Dominelli 2019). The definition of the protocols will be based on what has been observed by recent studies conducted on healthy people (Wuthrich et al., 2015; Schaer et al., 2018) and on patient populations in which respiratory dysfunction is a primary or secondary component of the pathology (Calcaterra et al., 2014; Pomidori et al., 2009). All planned interventions are safe and will be adapted to the obese patient.

DETAILED DESCRIPTION:
Project objectives are:

* evaluation of acute physiological responses, before and immediately after the single training session of the respiratory muscles conducted in the first days of hospitalization of the patients in the clinic.
* evaluation of physiological responses chronically, at the beginning and at the end of the three weeks of each workout The ultimate goal of this project will be to introduce targeted exercises for the respiratory muscles among the intervention guidelines for the prevention and reduction of obesity, especially juvenile, in order to break the vicious circle that is created in these patients, inactivity-obesity-inactivity, to create greater awareness of the body and the importance of a more active and healthy lifestyle and finally to have a greater consolidated effectiveness of intervention.

Materials and methods:

Subjects The study will be attended by 20 obese boys/young adults aged between 14 and 30 years old recruited at the Division of Auxology and the Division of Metabolic Diseases, Istitutio Auxologico Italiano, Piancavallo (VB).

Criteria for inclusion in the study group are:

1. BMI standard deviation score (SDS) > 2 for minors and BMI > 35 for patients aged > 18 years;
2. absence of structured physical activity programs (regular activity for more than 120 min/week) during the 6 months preceding the study;
3. absence of signs/symptoms referable to cardiovascular, respiratory, gastrointestinal, or musculoskeletal pathologies contraindicated for carrying out the tests.

Exercise protocol:

Upon entry into the clinic (PRE), immediately after the first respiratory training session (POST ACUTE) and at the end of the three weeks of hospitalization (POST CHRONIC), each subject will conduct the following exercise protocols on two experimental days separated by 48 hours on cycle ergometer:

1. incremental exercise (3 min rest, 30 watts for 3 minutes, 60 watts for 3 minutes, 90 watts for 3 minutes, with successive increments of 10 watts every minute) conducted until voluntary exhaustion
2. operation at constant load corresponding to 130% of the load corresponding to the gas exchange threshold (GET) conducted until voluntary exhaustion.

Measures:

The tests will be conducted under strict medical supervision, following standard safety protocols. All the measures and techniques proposed are non-invasive. The anthropometric characteristics (body circumferences and subcutaneous thickness at the thoracic and abdominal level) and the body composition of the patients will be determined by plicometry and tetrapolar impedancemetry at the beginning and at the end of the stay in the clinic.

* respiratory function and pulmonary gas exchange: spirometric indices, maximal voluntary ventilation at rest, pulmonary ventilation, breathing pattern (VT, fR, Ti/Ttot), PETO2 and PETCO2, pulmonary gas exchange measured "breath-by-breath" during exercise test (using a metabolimeter).
* V'O2peak and GET will be determined during incremental exercise, using standardized procedures (Salvadego et al. 2010).
* arterial saturation in O2 (SaO2) during exercise tests and during respiratory training sessions using finger pulsed oximetry.
* heart rate and heart rate variability during exercise tests and respiratory training sessions.
* spirometry (for evaluation of maximum lung capacity), to be performed in basal conditions and at the end of the protocol.
* perception of fatigue (using the Borg CR10 scale) during exercise tests.
* blood pressure, measured immediately before, during and immediately after exercise and immediately before and immediately after respiratory training sessions.

Respiratory muscle training protocol:

The recruited subjects will be randomly divided into two homogeneous groups in terms of number and basic characteristics of the subjects. A control group (CTRL) will carry out the standard integrated metabolic rehabilitation protocol with the addition of guided spontaneous breathing exercises lasting about 20 minutes per session for 12 sessions.

An experimental group (RMT) will carry out, in addition to the standard integrated metabolic rehabilitation protocol, a specific respiratory muscle training program according to the protocol recently proposed by Spengler et al. (Wuthrich et al., 2015; Schaer et al., 2018), adapted according to the baseline characteristics of the respiratory function of the subjects. The protocol includes 12 interval breathing training sessions, divided into 3 weeks (4 sessions/week) each lasting a total of about 12 minutes. Each respiratory training session includes 6 1-minute "sprint" breathing intervals followed by 1 minute of recovery. During the sprint intervals the subjects will breathe through a dedicated SpiroTiger instrument (Idiag AG, Fehraltorf, Switzerland) with the addition of a resistance (Schaer et al., 2018) which allows normocapnic hyperpnea against resistance. Subjects will be asked to breathe at a respiratory rate of 25-30 breaths/min with a constant tidal volume corresponding to approximately 60% of forced vital capacity. The target frequency will be adjusted on an individual basis and will be defined during the initial familiarization trials.

Expert staff will teach breathing exercises and follow patients during all training sessions.

ELIGIBILITY:
Inclusion Criteria:

* BMI standard deviation score (SDS) > 2 for patients aged < 18 years and BMI > 35 for patients aged > 18 years;
* absence of structured physical activity programs (regular activity for more than 120 min/week) during the 6 months preceding the study;
* absence of signs/symptoms referable to cardiovascular, respiratory, gastrointestinal, or musculoskeletal pathologies contraindicated for carrying out the tests.

Exclusion Criteria:

* presence of structured physical activity programs (regular activity for more than 120 min/week) during the 6 months preceding the study;
* presence of signs/symptoms referable to cardiovascular, respiratory, gastrointestinal, or musculoskeletal pathologies contraindicated for carrying out the tests.

Ages: 14 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
V'O2 peak during physical exercise protocol | Baseline and at the end of the training program (21 days)
  Change in V'O2 peak
Arterial saturation of O2 during physical exercise protocol | Baseline and at the end of the training program (21 days)
  Change in arterial saturation of O2

SECONDARY OUTCOMES:
Heart rate during physical exercise protocol | Baseline and at the end of the training program (21 days)
  Change in heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Site Piancavallo, Oggebbio, Verbania, Italy